CLINICAL TRIAL: NCT02133391
Title: Agency for Healthcare Research and Quality R18: Accountable Care Organizations (ACO)/ Public Health Collaborative Preventive Care Delivery to Priority Populations
Brief Title: Accountable Care Organizations/ Public Health Collaborative
Acronym: ACO/PH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-2395
Record Dates: First submitted 2013-12-16; First posted 2014-05-08 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Immunization Reminder System
Keywords: Accountable Care Organization; Comparative Effectiveness Research; Immunization/statistics & numerical data; Medicaid; Reminder Systems/economics; Reminder Systems/statistics & numerical data

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Practice-based reminder/recall or Usual care arm (Active Comparator): Practices participating in state immunization registry invited to reminder/recall (R/R) webinar trainings and provided educational materials to encourage immunization within their practices (child and adolescent trials only)
  Patients not randomized to the collaborative centralized R/R arm will receive usual care from their provider, which does not include R/R (adult trials only)
  Interventions: Other: Practice-based Reminder/Recall
- Collaborative centralized R/R (Experimental): Collaborative centralized reminder/recall (R/R) effort will be conducted by state immunization registry in collaboration with accountable care organizations and practices
  Interventions: Other: Centralized Reminder/Recall (R/R)

INTERVENTIONS:
Other: Centralized Reminder/Recall (R/R) — Method of increasing immunization delivery using reminder/recall techniques, which are implemented centrally.
  Arms: Collaborative centralized R/R
Other: Practice-based Reminder/Recall — Method of increasing immunization delivery using reminder/recall techniques, which are implemented at the practice level.
  Arms: Practice-based reminder/recall or Usual care arm

SUMMARY:
This study focuses on implementing and evaluating an evidence-based collaborative method of increasing immunization rates among preschool children, adolescents and adults within an Accountable Care Organization-Public Health collaborative. The infrastructure we will create through this project will serve as the framework for future collaborative delivery of other preventive services.

DETAILED DESCRIPTION:
The current project leverages newly formed Regional Care Collaborative Organizations (RCCO) in Colorado that are charged with providing comprehensive care for children and adults insured by Medicaid. With a new RCCO-public health collaborative we will implement a randomized controlled trial to test the effectiveness of 1) evidence-based collaborative centralized method of increasing immunization delivery using reminder/recall techniques versus 2) traditional practice-based reminder/recall techniques that are done by individual practices (not centrally) or usual care from their provider. These interventions have been previously developed by the study team in different clinical settings. The project will examine the collaborative centralized approach, implemented within the new RCCO-public health collaborative first among preschool children, the group in which it has been previously studied. We will then extend the method to new populations, including adolescents and adults within the RCCO and Denver Health (adults only), and will evaluate the effectiveness of the intervention in each population.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in Regional Care Collaborative Organizations (RCCOs) study practices in the regions covered by Colorado Access,
* Age 19-35 months,
* Age 11-17 years, or
* Age 18 years and older.
* Require an immunization according to Advisory Committee on Immunization Practices (ACIP) guidelines,
* Adult (18 and older) patients at 8 primary care sites who are enrolled in Denver Health and patients at 6 primary care RCCO study practices

Exclusion Criteria:

* Any child whose parents have requested removal from the immunization registry;
* Any adult who has requested removal from the immunization registry;
* Any child or adult with hypersensitivity to any component of one of the recommended vaccines;
* Any child or adult who has moved to a primary care provider other than one at the study practices.

Min Age: 19 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78354 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Vaccination Reminder/Recall | 2015-2017 (Year 2-4)
  1. Comparisons of receipt of any recommended vaccine and all recommended vaccines by study arm
  2. Comparisons of receipt of all needed vaccines
  3. Comparisons of receipt of specific targeted vaccines

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado School of Medicine, Children's Outcomes Research Program, Children's Hospital of Colorado
Locations (1):
- Children's Outcomes Research Program, University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurley LP, Beaty B, Lockhart S, Gurfinkel D, Dickinson LM, Roth H, Kempe A. Randomized controlled trial of centralized vaccine reminder/recall to improve adult vaccination rates in an accountable care organization setting. Prev Med Rep. 2019 May 22;15:100893. doi: 10.1016/j.pmedr.2019.100893. eCollection 2019 Sep. PMID 31193580
- [Derived] Hurley LP, Beaty B, Lockhart S, Gurfinkel D, Breslin K, Dickinson M, Whittington MD, Roth H, Kempe A. RCT of Centralized Vaccine Reminder/Recall for Adults. Am J Prev Med. 2018 Aug;55(2):231-239. doi: 10.1016/j.amepre.2018.04.022. Epub 2018 Jun 15. PMID 29910118